CLINICAL TRIAL: NCT04995328
Title: A Single Center, Open Label Clinical Investigation on the Treatment of Radiation Induced Dermatitis With Radiation Care® Gel
Brief Title: Clinical Investigation on the Treatment of Radiation Induced Dermatitis With Radiation Care® Gel
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: China Medical University Hospital (Other)
Responsible Party: Principal Investigator, Ying-Chun Lin, Attending Physician, Division of Radiation Oncology, Principal Investigator, China Medical University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: CMUH110-REC1-122
Record Dates: First submitted 2021-07-21; First posted 2021-08-06 (Actual); Last update posted 2023-09-06 (Actual); Status verified 2023-09

CONDITIONS: Radiation Dermatitis
Keywords: Lonicera japonica; breast cancer; head and neck cancer
MeSH Terms: conditions — Radiodermatitis; Breast Neoplasms; Head and Neck Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Radiation Care Gel application (Experimental): Radiation Care® gel is instructed to use on the target skin area accepted radiation therapy twice daily.
  Interventions: Other: Radiation Care Gel

INTERVENTIONS:
Other: Radiation Care Gel — The investigational medical product of this study is a hydrogel, Radiation Care® gel which increases moisturizing and it can be applied to the target areas including skin folds and creases.

SUMMARY:
The radiotherapy after surgery reduces the risk of recurrence and death is widely used for standard treatment for cancer including breast cancer and head and neck cancer. However, radiation dermatitis is a common side effect and major adverse event of radiotherapy. Radiation induces skin inflammation resulting in redness, itchiness and peeling skin. Radiation dermatitis may be acute or chronic. Acute skin changes occur within 90 days of initiating therapy due to inflammation and DNA damage and chronic skin changes may occur after several weeks or years. Radiation-irritated skin is a treatment-induced symptom caused by radiation dose-limiting toxicity. It damages skin structure and causes a variety of symptoms of cuticle thinning, reducing of collagen in subcutaneous, sweat glands damage, sebaceous glands damage and basal membrane damage. These conditions lead patients to lost work productivity, wound care costs, social isolation, altered body image and affect a patient's quality of life and mental health both during and after treatment and even interrupts the treatment schedule.

The treatment of radiation dermatitis is an essential component of radiotherapy. The common treatment includes agents and other dressing products, such as corticosteroid cream, hyaluronic acid, aloe and sucralfate, which are used to prevent or reduce severity of dermatitis. But there is no clear therapeutic or nursing guideline supporting continuous treatment of radiation dermatitis by topical agents currently.

In this study, Radiation Care® gel which contain Japanese honeysuckle extract will be used in breast and head and neck cancer patients to test the safety and efficacy to prevent radiation dermatitis and alleviate their radiation-irritated skin symptoms.

The primary objective of this study is to evaluate the clinical outcomes of "Radiation Care" gel application in breast cancer and head and neck cancer patients who have radiation dermatitis or radiation-irritated skin due to the radiotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Participants must be males or non-pregnant or non-lactating females at least 20 years of age.
* Subject must meet one of the following conditions:

  1. Diagnosis of non-inflammatory breast adenocarcinoma or in situ breast cancer which were treated by operation with or without adjuvant or neoadjuvant hormonal treatment.
  2. Diagnosis of epithelial carcinoma of nasopharynx, oropharynx, oral cavity, larynx, hypopharynx, paranasal sinus and salivary glands which were treated with or without operation, concurrent chemotherapy is accepted, in head and neck cancer patients.
* Patients were scheduled to receive at least three sessions of radiotherapy per week (1 session per day) for at least five weeks using standard irradiation fraction (with at least 1.8 Gy per session) for total dose of at least 50 Gy.
* Participant willing and must give signed informed consent.

Exclusion Criteria:

* Prior breast reconstructions, implants, and/or expanders.
* Previous radiotherapy to the area to be treated with radiation therapy (head and neck area or breast and thorax areas).
* Concurrent chemotherapy in breast cancer patients.
* Concurrent targeted therapy in head and neck cancer patients.
* Known radiosensitivity syndromes (e.g. Ataxia-telangiectasia)
* Collagen vascular disease, vasculitis, unhealed surgical sites, breast infections, rashes or unhealed wounds in the radiation field or systemic lupus erythematosus (SLE).
* Systemic diseases known to delay the skin healing process such as diabetes mellitus or severe renal failure.
* Use of a tissue-equivalent bolus.
* Use of over-the-counter topical medications containing steroids.
* Participation in any clinical trial in the prior 30 days from baseline.
* Any condition that, in the judgement of the investigator could impose hazards to the patient if study therapy is initiated or affect the participation of the patient in the study.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2021-08-03 (Actual); Primary Completion 2022-08-26 (Actual); Study Completion 2022-10-07 (Actual)

PRIMARY OUTCOMES:
To observe the proportion of patients with grade 2 radiation dermatitis (according to CTCAE) at week 5. | at 5 weeks
  According to Common Terminology Criteria for Adverse Events (CTCAE) system by national cancer institute, radiation induced skin toxicities is scored in severity in the following grades:
  Grade 1: faint erythema or dry desquamation Grade 2: moderate to brisk erythema; moist desquamation confined to skin folds; moderate edema Grade 3: moist desquamation in areas other than skin folds and creases; bleeding induced by minor trauma or abrasion Grade 4: skin necrosis or large ulcerations; spontaneous bleeding or require surgical procedures Grade 5: with lethal consequences

SECONDARY OUTCOMES:
To evaluate radiation-irritated situation after 3 months of Radiation Care® gel application in breast cancer and head and neck cancer patients who completed the post-operative radiotherapy. | Day0 (baseline), 1-Week, 2-Week, 3-Week, 4-Week, 5-Week, 6-Week, 7-Week, Post-radiotherapy 2-week, Post-radiotherapy 6-week
  The skin condition of target area will be observed and recorded at clinical visit. The measurement include:
  1. Erythema grade:
     Grade 1: Very faint erythema: Skin has a very light pink color. Grade 2: Faint erythema: Skin reaction is more apparent with clear borders but is still pink with more intensity.
     Grade 3: Bright erythema: Erythema is apparent in bright pink and borders are clearly defined.
     Grade 4: Very bright erythema: Skin is bright red, borders are very well defined, capillaries and bruising may be visible.
  2. Graded according to CTCAE rate
  3. Moisture percentage will be detected by MoistureMeter SC
To compare the moisture percentage at the radiotherapy site from baseline to follow-up visit. | Up to 12-13 weeks (depend on different times of radiotherapy in breast cancer and head and neck cancer): From Day0 (baseline) to 2-Week, 4-Week, 6-Week, Post-radiotherapy 2-week, Post-radiotherapy 6-week (End of study)
  Moisture percentage will be detected by MoistureMeter SC for every two weeks.
The score of quality of life with the Skindex-16 questionnaire performed every two weeks. | Up to 12-13 weeks (depend on different times of radiotherapy in breast cancer and head and neck cancer): From Day0 (baseline) to 2-Week, 4-Week, 6-Week, Post-radiotherapy 2-week, Post-radiotherapy 6-week (End of study)
  The Skindex-16 is an assessment using numerical analog scales (0 = never bothered to 6 = always bothered), used to comprehensively measure the effects of skin diseases on subject's quality of life including burden of symptoms, social function and emotional state that the CTCAE does not take into account. The higher scores present poorer quality of life.

CONTACTS AND LOCATIONS:
Locations (1):
- China Medical University Hospital, Taichung, Taiwan

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Ahn S, Sung K, Kim HJ, Choi YE, Lee YK, Kim JS, Lee SK, Roh JY. Reducing Radiation Dermatitis Using a Film-forming Silicone Gel During Breast Radiotherapy: A Pilot Randomized-controlled Trial. In Vivo. 2020 Jan-Feb;34(1):413-422. doi: 10.21873/invivo.11790. PMID 31882508
- [Background] Clemenson C, Liu W, Bricout D, Soyez-Herkert L, Chargari C, Mondini M, Haddad R, Wang-Zhang X, Benel L, Bloy C, Deutsch E. Preventing Radiation-Induced Injury by Topical Application of an Amifostine Metabolite-Loaded Thermogel. Int J Radiat Oncol Biol Phys. 2019 Aug 1;104(5):1141-1152. doi: 10.1016/j.ijrobp.2019.04.031. Epub 2019 May 4. PMID 31063799
- [Background] Wang L, Jiang Q, Hu J, Zhang Y, Li J. Research Progress on Chemical Constituents of Lonicerae japonicae flos. Biomed Res Int. 2016;2016:8968940. doi: 10.1155/2016/8968940. Epub 2016 Jun 14. PMID 27403439
- [Background] Jeong YT, Jeong SC, Hwang JS, Kim JH. Modulation effects of sweroside isolated from the Lonicera japonica on melanin synthesis. Chem Biol Interact. 2015 Aug 5;238:33-9. doi: 10.1016/j.cbi.2015.05.022. Epub 2015 Jun 5. PMID 26051519
- [Background] Wu L. Effect of chlorogenic acid on antioxidant activity of Flos Lonicerae extracts. J Zhejiang Univ Sci B. 2007 Sep;8(9):673-9. doi: 10.1631/jzus.2007.B0673. PMID 17726749
- [Background] Liao Y, Dong S, Kiyama R, Cai P, Liu L, Shen H. Flos lonicerae extracts and chlorogenic acid protect human umbilical vein endothelial cells from the toxic damage of perfluorooctane sulphonate. Inflammation. 2013 Jun;36(3):767-79. doi: 10.1007/s10753-013-9603-5. PMID 23392856